CLINICAL TRIAL: NCT05276544
Title: The Effect of Telephone and Video Counseling Given to Obese Individuals on Weight Loss and Quality of Life in the COVID-19 Pandemic: an RCT
Brief Title: The Effect of Telephone and Video Counseling on Weight Loss and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Collaborators: Amasya University (Other)
Responsible Party: Principal Investigator, ümüş özbey yücel, Clinical Researcher of the Amasya University Nutrition and Diet Department, Ankara University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AmasyaUniv
Record Dates: First submitted 2022-03-03; First posted 2022-03-11 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Weight Loss; Obesity
Keywords: Obesity; Weight Loss; COVID-19 pandemic
MeSH Terms: conditions — Weight Loss; Obesity; COVID-19 | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- phone counseling (Experimental): dietary intervention via phone counseling
  Interventions: Behavioral: Dietary intervention
- video counseling (Experimental): dietary intervention via video counseling
  Interventions: Behavioral: Dietary intervention
- Traditional follow up (Experimental): dietary intervention via traditional follow up
  Interventions: Behavioral: Dietary intervention

INTERVENTIONS:
Behavioral: Dietary intervention — Dietary intervention: Preparation and follow-up of diet program.

SUMMARY:
Individuals with obesity are at higher risk for severe disease, hospitalizations, and death from the SARS-CoV-2 virus. Social distancing guidelines intended to prevent viral spread during the COVID-19 pandemic resulted in major changes to daily routines . Several studies have demonstrated that individuals with overweight/obesity reported worsening mental health, poor eating habits , less physical activity (PA) since the onset of the COVID-19 pandemic. Because of these pandemic rules, the use of phone/video consultancy applications and online classes for body weight control and diet monitoring is increasing. Therefore, in this study it is aimed to determine the effect of diet counseling via phone or video on weight loss and to compare it with the traditional follow-up method in the COVID-19 pandemic.

DETAILED DESCRIPTION:
The use of phone/video consultancy applications for body weight control and diet monitoring is increasing. One of the main reasons for this situation is that individuals care more about the social distance rule as a result of the increase in health concerns after the COVID-19 (SARS-CoV-2) pandemic. In addition, due to the uncertainty of how long the pandemic will last, many people are adapting to online applications and programs quicly. However, it's unclear which method of phone/video-based diet counseling is more successful or preferable to traditional diet follow-up. Based on the above-mentioned information; in this study, it is aimed to determine the effect of diet counseling via phone or video on weight loss and to compare it with the traditional follow-up method in the COVID-19 pandemic.

Individuals who meet the research criteria will randomize according to their file numbers (with the ramdomizer program) and divide into 3 groups: telephone counseling (15), video counseling (15) and traditional follow-up group (Figure 1.). Food consumption records, anthropometric measurements and quality of life scale scores of all individuals will record at the beginning and end of the study (Figure 2.). In order to prevent interaction between individuals, all diet programs will prepare at different times and individually.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 20-65
* Being obese (BMI≥30 kg/m2)
* Having a smartphone with internet access and being competent to use it
* Volunteering to participate in research

Exclusion Criteria:

* Being pregnant/lactating
* Having a hearing problem
* Being on a followed diet program

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-18 (Actual)

PRIMARY OUTCOMES:
Weight chance | At the end of the 3 months
  BMI (kilogram/ metre2 (kg/m2))

SECONDARY OUTCOMES:
Quality of Life Score | At the end of the 3 months
  The score ranges from 0 to 100 points, with an increased score reflecting improved quality of life

CONTACTS AND LOCATIONS:
Overall Officials: ümüş Ö yücel, Dr, Principal Investigator — Ankara University
Locations (1):
- Ümüş Özbey, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No